Official Title: A Pilot Study Evaluating Pemetrexed in ECOG Performance Status 3

Patients With Stage IV Non-squamous Non-small Cell Lung Cancer

NCT02426658

IRB-Approved Date: 3/21/2018



Section of Hematology and Oncology

# A PILOT STUDY EVALUATING PEMETREXED IN ECOG PERFORMANCE STATUS 3 PATIENTS WITH STAGE IV NON-SQUAMOUS NON-SMALL CELL LUNG CANCER

Informed Consent Form to Participate in Research Stefan C. Grant, MD, JD, MBA, Principal Investigator

#### Introduction

You are invited to be in a research study. Research studies are designed to gain scientific knowledge that may help other people in the future. You are being asked to take part in this study because you have Stage IV non-small cell lung cancer. Your participation is voluntary. Please take your time in making your decision as to whether or not you wish to participate. Ask your study doctor or the study staff to explain any words or information contained in this informed consent document that you do not understand. You may also discuss the study with your friends and family.

#### WHY IS THIS STUDY BEING DONE?

The purpose of this research study is to see what effects (good and bad) the chemotherapy drug pemetrexed has on you and your condition. Pemetrexed has been approved by the US Food and Drug Administration (FDA) for patients with advanced lung cancer, but current cancer treatment guidelines limit chemotherapy use to patients who are ambulatory and capable of all self-care. Pemetrexed has shown anti-cancer benefit and been well-tolerated in these patients. Side effects can be minimized with folic acid, vitamin B12, and corticosteroids. In addition to these patients, we believe that pemetrexed can provide anti-cancer benefit and be well-tolerated in patients who are capable of only limited self-care.

# HOW MANY PEOPLE WILL TAKE PART IN THE STUDY?

We anticipate that 30 people will take part in this study.

### WHAT IS INVOLVED IN THE STUDY?

Prior to beginning the study, we will collect information on your demographics, medical history, current medications, physical functioning, quality of life, height, weight, and vital signs. We will need to draw blood to check your blood counts and to test for pregnancy in women of childbearing potential. You will also have a CT scan to take tumor measurements.

Prior to each treatment we will check your blood counts. At each treatment we will check your vital signs and collect information about your physical functioning and quality of life.


Adult Consent Form

Version: 03-04-15



Pemetrexed will be given as an intravenous infusion on the first day of each 21-day treatment cycle. To help prevent and reduce treatment side effects, you will be given folic acid, vitamin B12, and a corticosteroid. You will start taking folic acid once daily at least 7 days before the first dose of pemetrexed. You will continue taking folic acid during the full course of therapy and for 21 days after the last dose of pemetrexed. In addition to this, you will receive an intramuscular injection of vitamin B12 at least 1 week prior to the first dose of pemetrexed and at least every 3 cycles thereafter. Dexamethasone is an oral corticosteroid that you will take twice daily the day before, the day of, and the day after pemetrexed administration.

You will have a CT scan every 6 weeks to assess the effectiveness of the pemetrexed treatment on the tumor

You will have approximately 1 teaspoon of blood withdrawn from a vein before starting the study and then 1 teaspoon during each treatment cycle. The total amount of blood withdrawn during the study will be depend on how many treatment cycles you participate in this study.

#### HOW LONG WILL I BE IN THE STUDY?

You may continue with the study treatment until you decide to withdraw from the study or your condition changes in such a way that your physician does not think you should continue on this study.

You can stop participating at any time. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff first to learn about any potential health or safety consequences.

#### WHAT ARE THE RISKS OF THE STUDY?

Being in this study involves some risk to you. You should discuss the risk of being in this study with the study staff. The most common side effects of treatment with Pemetrexed are fatigue, nausea, and anorexia. Other less common side effects include a low red blood cell count, low platelet count, low white blood cell count, mouth sores, diarrhea, and stomach irritation.

There also may be other side effects that we cannot predict. You should tell the research staff about all the medications, vitamins and supplements you take and any medical conditions you have. This may help avoid side effects, interactions and other risks.

In addition, there is a slight risk of a breach of confidentiality. We will do our best to protect your confidential information. Taking part in this research study may involve providing information that you consider confidential or private. Efforts, such as coding research records, keeping research records secure and allowing only authorized people to have access to research records, will be made to keep your information safe.

You may experience discomfort, bruising and/or bleeding where the needle is inserted when you have blood drawn. Occasionally some people become dizzy lightheaded or feel faint. Infection may occur on rare occasions. Frequent donation of blood can result in low iron in your blood


Adult Consent Form

Version: 03-04-15



(iron deficient anemia).

# Reproductive Risks and other Issues to Participating in Research

Due to unknown risks and potential harm to the unborn fetus, sexually active women of childbearing potential must use a reliable method of birth control while participating in this study. Reliable methods of birth control are: abstinence (not having sex), oral contraceptives, intrauterine device (IUD), Depo-Provera, tubal ligation, or vasectomy of the partner (with confirmed negative sperm counts) in a monogamous relationship (same partner). An acceptable, although less reliable, method involves the careful use of condoms and spermicidal foam or gel and/or a cervical cap or sponge. We encourage you to discuss this issue further with your physicians if you have any questions.

Pregnant women are excluded from participation in this study. Because some methods of birth control are not 100% reliable, a pregnancy test is required at least 10 days from your last normal menstrual period, if you are a sexually active woman of childbearing potential.

#### ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

If you agree to take part in this study, there may or may not be direct benefit to you. Based on experience with Pemetrexed in more physically active patients with lung cancer, researchers believe it may be of benefit to patients like you. Because individuals respond differently to therapy, no one can know in advance if it will be helpful in your particular case. In addition, we hope the information learned from this study will benefit other people in the future.

#### WHAT OTHER CHOICES ARE THERE?

You do not have to be in this study to receive treatment. You should talk to your doctor about all the choices you have. Instead of being in this study, you have these options: Another clinical trial, best supportive care.

## What About My Health Information?

In this research study, any new information we collect from you and/or information we get from your medical records or other facilities about your health or behaviors is considered <u>Protected Health Information</u>. The information we will collect for this research study includes:

Demographics, medical history, current medications, physical exam details, vital signs, height, weight, performance status, tumor measurements, bloodwork (Complete Blood Count (CBC), serum chemistry), treatment-related side effects or symptoms.

If this research study involves the diagnosis or treatment of a medical condition, then Protected Health Information collected from you during this study will be placed in your medical record, and may be used to help treat you, arrange payment for your care, or assist with Medical Center operations.

We will make every effort to keep your Protected Health Information private. We will store records of your Protected Health Information in a cabinet in a locked office or on a password


Adult Consent Form

Version: 03-04-15



protected computer. Only the following people or organizations will be granted access to your Protected Health Information:

- 1) The study investigator and his/her staff, or others at Wake Forest University Health Sciences who oversee research
- 2) Other people or laboratories providing services for this research project on behalf of Wake Forest University Health Sciences and Wake Forest University Baptist Medical Center

If required by law or court order, we might also have to share your Protected Health Information with a judge, law enforcement officer, government agencies, or others. If your Protected Health Information is shared with any of these groups it may no longer be protected by federal or state privacy rules.

Any Protected Health Information collected from you in this study that is maintained in the research records will be kept for an indeterminate period of time. This authorization does not expire. Any research information entered into your medical record will be kept for as long as your medical record is kept by the Medical Center. You will not be able to obtain a copy of your Protected Health Information in the research records until all activities in the study are completely finished.

You can tell Dr. Stefan Grant that you want to take away your permission to use and share your Protected Health Information at any time by sending a letter to this address:



However, if you take away permission to use your Protected Health Information you will not be able to be in the study any longer. We will stop collecting any more information about you, but any information we have already collected can still be used for the purposes of the research study.

By signing this form you give us permission to use your Protected Health Information for this study.

If you choose to participate in this study, your medical record at Wake Forest University Baptist Medical Center will indicate that you are enrolled in a clinical trial. Information about the research and any medications or devices you are being given as a participant may also be included in your medical record. This part of the medical record will only be available to people who have authorized access to your medical record. If you are not a patient at this Medical Center, a medical record will be created for you anyway to ensure that this important information


Adult Consent Form

Version: 03-04-15



is available to doctors in case of an emergency.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this Web site at any time.

Laboratory test results and other medical reports created as a result of your participation in the research study may be entered into the computer systems of Wake Forest University Health Sciences and North Carolina Baptist Hospital. These will be kept secure, with access to this information limited to individuals with proper authority, but who may not be directly involved with this research study.

#### WHAT ARE THE COSTS?

Taking part in this study may lead to added costs to you or your insurance company. We will give you an estimate of what the added cost may be based on your particular situation and insurance coverage.

#### WILL YOU BE PAID FOR PARTICIPATING?

You will receive no payment or other compensation for taking part in this study.

Parking validation will be provided for study-related visits.

The findings from this research may result in the future development of products that are of commercial value. There are no plans to provide you with financial compensation or for you to share in any profits if this should occur.

#### WHO IS SPONSORING THIS STUDY?

This study is being sponsored by the Comprehensive Cancer Center of Wake Forest University. The sponsor is providing money or other support to Wake Forest University Health Sciences to help conduct this study. The researchers do not, however, hold a direct financial interest in the sponsor or the product being studied.

# WHAT HAPPENS IF YOU EXPERIENCE AN INJURY OR ILLNESS AS A RESULT OF PARTICIPATING IN THIS STUDY?

Should you experience a physical injury or illness as a direct result of your participation in this study, Wake Forest University School of Medicine maintains limited research insurance coverage for the usual and customary medical fees for reasonable and necessary treatment of such injuries or illnesses. To the extent research insurance coverage is available under this policy the reasonable costs of these necessary medical services will be paid, up to a maximum of \$25,000. Wake Forest University Baptist Medical Center holds the insurance policy for this coverage. It provides a maximum of \$25,000 coverage for each claim and is limited to a total of \$250,000 for all claims in any one year. The Wake Forest University School of Medicine, and the North Carolina Baptist Hospitals, Incorporated do not assume responsibility to pay for these medical services or to provide any other compensation for such injury or illness. Additional


Adult Consent Form

Version: 03-04-15



information may be obtained from the Medical Center's Director of Risk and Insurance Management, at

If you are injured, the insurer may require information such as your name, social security number, and date of birth in order to pay for your care. This is because the insurer is required by law to report any payments made to cover the care of any persons who are members of a government insurance plan to the Department of Health and Human Services.

You do not give up any legal rights as a research participant by signing this consent form. For more information on medical treatment for research related injuries or to report a study related illness, adverse event, or injury you should call Dr. Stefan Grant at

#### WHAT ARE MY RIGHTS AS A RESEARCH STUDY PARTICIPANT?

Taking part in this study is voluntary. You may choose not to take part or you may leave the study at any time. Refusing to participate or leaving the study will not result in any penalty or loss of benefits to which you are entitled. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff first to learn about any potential health or safety consequences. The investigators also have the right to stop your participation in the study at any time. This could be because it is in your best medical interest, your condition worsened, new information becomes available, you had an unexpected reaction, you failed to follow instructions, or because the entire study has been stopped.

You will be given any new information we become aware of that would affect your willingness to continue to participate in the study.

# WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?

For questions about the study or in the event of a research-related injury, contact the study investigator, Dr. Stefan Grant, at

The Institutional Review Board (IRB) is a group of people who review the research to protect your rights. If you have a question about your rights as a research participant, or you would like to discuss problems or concerns, have questions or want to offer input, or you want to obtain additional information, you should contact the Chairman of the IRB at

You will be given a copy of this signed consent form.

#### **SIGNATURES**

I agree to take part in this study. I authorize the use and disclosure of my health information as described in this consent and authorization form. If I have not already received a copy of the Privacy Notice, I may request one or one will be made available to me. I have had a chance to ask questions about being in this study and have those questions answered. By signing this


Adult Consent Form

Version: 03-04-15



consent and authorization form, I am not releasing or agreeing to release the investigator, the sponsor, the institution or its agents from liability for negligence.

| Subject Name (Printed): | | | |
|---------------------------|-------|-------|-------|
| Subject Signature: | Date: | Time: | am pm |
| Person Obtaining Consent: | Date: | Time: | am pm |

 Adult Consent Form

Version: 03-04-15